CLINICAL TRIAL: NCT05985343
Title: The Impact of Sugammadex on Ileus After Abdominal Wall Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clayton Petro (Other)
Responsible Party: Sponsor-Investigator, Clayton Petro, Assistant Professor of Surgery Lerner College of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-700
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Hernia, Ventral; Ileus
MeSH Terms: conditions — Hernia, Ventral; Ileus | interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to receive sugammadex or neostigmine/glycopyrrolate for reversal of neuromuscular blockade
Who Masked: Participant
Masking Description: The patient will be blinded as to what medication they receive for reversal of neuromuscular blockade
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine/Glycopyrrolate (Other): Patients assigned to the control arm receive the standardized reversal neostigmine dose with on-label dosing (0.03-0.07mg/kg) and a fixed ratio of glycopyrrolate
  Interventions: Drug: Neostigmine / Glycopyrrolate
- Sugammadex (Other): Patients randomized to the experimental arm will receive an IV dose of sugammadex according to the package insert of 2 mg/kg for ≥ 2 twitches, 4 mg/kg for 1-2 post-tetanic twitches
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine / Glycopyrrolate — Patients will receive standard of care for reversal of neuromuscular blockade
  Other Names: Control arm
  Arms: Neostigmine/Glycopyrrolate
Drug: Sugammadex — Patients will receive sugammadex for reversal of neuromuscular blockade
  Other Names: Experimental arm
  Arms: Sugammadex

SUMMARY:
The aim of the study is to determine if the usage of sugammadex would reduce the time to return of bowel function when compared to standard of care (neostigmine/glycopyrrolate) when used for neuromuscular blockade reversal in patients with open abdominal wall reconstruction (AWR).

DETAILED DESCRIPTION:
The investigators baseline postoperative ileus (POI) rate in the setting of open abdominal wall reconstruction (AWR) is similar to patients undergoing an open bowel resection and often prolongs patients' hospital stay. Therefore, the investigators aim to determine whether the use of sugammadex has a clinically significant impact on return of postoperative bowel function and prevention of POI in these patients.

The primary outcome is GI-2: postoperative time until passage of 1st bowel movement and tolerance of solid food.

The investigators hypothesize:

* postoperative time to return of bowel function (GI-2) after open AWR will be significantly shorter for patients who receive sugammadex for reversal of neuromuscular blockade when compared to those receiving standard of care (neostigmine/glycopyrrolate).
* patients who receive sugammadex for reversal of neuromuscular blockade will have a reduced incidence of POI requiring nasogastric tube (NG) placement, and decreased length of hospital stay when compared to standard of care.

Specific Aim 1: To determine if the use of sugammadex for neuromuscular blockade reversal reduces the time to postoperative GI-2 bowel function compared to neostigmine/glycopyrrolate for neuromuscular blockade reversal.

Specific Aim 2: To determine if sugammadex reduces the incidence of postoperative NG placement compared to neostigmine/glycopyrrolate for neuromuscular blockade reversal.

Specific Aim 3: To determine if sugammadex reduces postoperative length of stay following AWR compared to neostigmine/glycopyrrolate for neuromuscular blockade reversal.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old
* Patients requiring an open ventral hernia repair with retromuscular mesh placement and at least one myofascial advancement flap
* Hernias with fascial defects < 20cm wide
* Non-emergent cases

Exclusion Criteria:

* Known serious or severe hypersensitivity reaction to sugammadex or any of the ingredients in sugammadex.
* Hernias with fascial defects > 20cm wide
* Concomitant treatment with a strong or moderate cytochrome P450 3A4 inhibitor (e.g., Ketoconazole and other anti-fungals, Clarithromycin, HIV protease inhibitors, diltiazem, erythromycin, verapamil) or strong CYP3A4 inducers (e.g., rifampin).
* Known small bowel obstruction (SBO) at the time of hernia repair
* Suspected SBO or at risk of recurrent SBO at the time of hernia repair - at the discretion of the staff surgeon.
* Nasogastric (NG), orogastric (OG), or gastric (eg. PEG) in place at the time of hernia repair and left in beyond the morning of the first postoperative day.
* Patients with a stoma.
* Cancer with increased risk of gastro-duodenal perforation (e.g., infiltrative gastrointestinal tract malignancy, recent gastrointestinal tract surgery, diverticular disease including diverticulitis, ischemic colitis, or concomitantly treated with bevacizumab) - at the discretion of the staff surgeon.
* Disorder that could alter the integrity of the gastrointestinal lining (e.g., Crohn's disease) - at the discretion of the staff surgeon.
* Severe hepatic failure (Child-Pugh Class C).
* Clinically relevant hepatic failure (e.g. cirrhosis) - at the discretion of the staff surgeon.
* Severe renal failure (GFR<30ml/min, on dialysis, or have an arteriovenous fistula, indwelling hemodialysis catheter or peritoneal dialysis catheter) - at the discretion of the staff surgeon.
* Pregnant or planning to become pregnant during study period.
* Breastfeeding or planning to breastfeed during study period.
* Clinically relevant alteration of the blood-brain-barrier - at the discretion of the staff surgeon.
* Other contraindication to sugammadex as documented by a physician.
* Unable to give informed consent; vulnerable populations; non-English speaking.
* Emergent operation.
* Undergoing minimally invasive approaches.
* Undergoing repair with mesh placed in a position other than retromuscular.
* Chronic opioid users, as defined by the daily use of opioids for at least 90 days within the past year
* Inability to safely extubate the patient at the end of the surgery for any reason, as determined by the operative team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Time to GI-2 bowel function after surgery | From time of randomization to progression of bowel function, which is an average of 87 hours, or until 1 month after randomization; whichever comes first
  The median time to first postoperative bowel movement and tolerance of solid food (defined as GastroIntestinal-2), as measured in hours, will be recorded for each patient and compared between the two groups.

SECONDARY OUTCOMES:
Length of stay | From time of randomization to progression allowing safe discharge home, which is an average of 6 days, or until 1 month after randomization; whichever comes first
  Duration of hospital stay as measured in hours from end of surgery to placement of discharge order will be
Postoperative nasogastric tube placement rate | Up to 1 month after randomization
  Placement of nasogastric tube for nausea/vomiting after surgery will be recorded and compared between the two groups.
Postoperative complications | Up to 1 month after randomization
  All postoperative complications will be recorded and compared between the two groups
Postoperative pain | Postop day 1, 2, 3, and 4
  Postop pain will be assessed using the Pain Numeric Rating Scale (NRS-11) where patients will report their pain on a 0-10 scale, where higher scores mean worse pain. Overall scores will be compared between the two groups.
Opioid used in morphine milligram equivalents | Postop day 1, 2, 3, and 4
  Total postoperative opioid use will be recorded after converted into morphine milligram equivalents (MMEs) and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton C Petro, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Abdominal Core Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No